CLINICAL TRIAL: NCT04827017
Title: Acute and Chronic Pulmonary and Renal Complications Following Contractiong Coronavirus Severe Respiratory Distress Syndrome.
Brief Title: Acute and Chronic Pulmonary and Renal Complications Following Contracting Severe Respiratory Distress Syndrome Coronavirus-19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mina Maher, Lecturer of anesthesia and ICU, Minia University
Other Study IDs: 278/3-2021
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Pulmonary and Renal State

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: follow up — follow up population

SUMMARY:
Tracking post- corona virus infection pulmonary and renal complications

DETAILED DESCRIPTION:
Mortality from pulmonary and renal system is highly noticable with COVID-19 pandemic . We trying to monitor compliction

ELIGIBILITY:
Inclusion Criteria:

* All COVID 19 patients admitted to ICU

Exclusion Criteria:

* Refusal to participate

Ages: 20 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All COVID positive population
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-04-05 (Estimated); Primary Completion 2021-07-05 (Estimated); Study Completion 2021-07-10 (Estimated)

PRIMARY OUTCOMES:
renal function | 12 weeks
  serum creatinine